CLINICAL TRIAL: NCT02736929
Title: The Effect of Reducing Posttraumatic Stress Disorder Symptoms on Cardiovascular Risk
Acronym: ACCEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00067912
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Processing Therapy - Cognitive (Active Comparator): Cognitive Processing Therapy - Cognitive (CPT-C), is a brief cognitive behavioral treatment for PTSD. CPT-C consists of 2 hours of therapy each week for 6 weeks (i.e., two sessions).
  Interventions: Behavioral: Cognitive Processing Therapy - Cognitive
- Waiting Period Control (WP-CON) (No Intervention): WP-CON group will receive minimal attention in the form of weekly telephone calls to assess current emotional state and to provide supportive, nondirective, brief counseling if participants report experiencing a crisis. Any participant assigned to the WP-CON group will be given the opportunity to receive CPT-C after the post-waiting period assessment.

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy - Cognitive — CPT-C is a brief cognitive behavioral treatment for PTSD. It consists of 2 hours of therapy each week for 6 weeks (i.e., two sessions).
  Other Names: CPT-C
  Arms: Cognitive Processing Therapy - Cognitive

SUMMARY:
Some individuals who are exposed to traumatic events experience both psychological and cardiovascular changes that affect their health and well-being. The purpose of this study is to learn more about how reducing the psychological symptoms (such as those that occur with posttraumatic stress disorder, or PTSD) affects cardiovascular systems that regulate heart and blood pressure.

DETAILED DESCRIPTION:
There is a fundamental gap in the understanding of how a diagnosis of post-traumatic stress disorder (PTSD) portends excess risk of coronary heart disease (CHD). This is primarily because of two reasons: (1) the core studies which provide support for an association between PTSD and CHD risk depended on lengthy follow-up periods with no repeat measurement of either PTSD or other related cardiovascular risk factors; (2) PTSD is highly comorbid with both adverse health behaviors and with psychiatric comorbidity that also vary across time and could largely explain the association between PTSD and increased risk of CHD. The long-term goal is to better understand whether there is a direct link between PTSD and CHD risk, as well as to ascertain the role of candidate pathophysiological mechanisms. The study proposed in this application is designed to examine how changes in PTSD symptoms following an established therapeutic intervention (Cognitive Processing Therapy) affect CHD disease pathways in individuals with PTSD. This design will permit an evaluation of the hypothesis that individuals who show significant improvement in PTSD symptoms will also show improvement in CHD risk biomarkers, and individuals who fail to show improvement or show worsening PTSD symptoms, will show no change or worsening in CHD biomarker activity. The study will also provide an evaluation of the role of key stress-related CHD biomarkers as mechanisms underlying the increased CHD risk burden associated with PTSD. Choice of CHD biomarkers focused on the established association of PTSD with chronic activation of stress response systems and includes autonomic nervous system dysregulation, chronic systemic inflammation, and vascular endothelial dysfunction. The proposed research is significant because it is expected to provide knowledge of the role of both the direct impact of PTSD symptoms on CHD risk pathways and the role of these systems as candidate mechanisms underlying the relationship between PTSD and CHD risk. By better defining how PTSD is a risk factor for CHD, as well as identifying the disease pathways involved, the proposed study will help inform strategies for CHD prevention, as well as guide optimal medical management for vulnerable men and women with PTSD, especially in those who refrain or who are refractory to psychiatric treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 40 and 65;
* Has current PTSD lasting at least three months, based on the Clinician Administered PTSD Scale (CAPS), DSM 5 version, with a CAPS total score of 25 or greater; and
* Will have been stable on any current psychiatric medications for four weeks prior to the Time 1 assessment.

Exclusion Criteria:

* Is currently participating in evidence-based trauma focused therapy (e.g., CPT, prolonged exposure) for PTSD (current or past 6 months);
* Has current dementia or other memory loss condition, as indicated by self-report or as indicated by scores less than 20 on the Montreal Cognitive Assessment (MoCA);
* Has current psychotic spectrum disorder or bipolar disorder;
* Has current uncontrolled substance use disorder that would interfere with his/her ability to perform study procedures;
* Has a urine drug screen positive for cocaine and/or methamphetamine and reports regular use of that substance;
* Has severely impaired hearing or speech;
* Is pregnant;
* Has established heart disease, abnormal heart rhythm, advanced cancer, or epilepsy
* Has HIV positive status with unstable disease status and/or unstable medication use;
* Has current exposure to ongoing trauma (e.g., physically abusive relationship);
* Has prominent suicidal or homicidal ideation (as assessed through a clinical interview);
* Has a serious/terminal illness or other health problem that would prohibit participation in the study;
* Has an inflammatory condition such as infection, fever, one-month history of accident or surgery, rheumatoid arthritis, lupus, or inflammatory bowel disease.
* Is unwilling to accept randomization; or
* Cannot agree to attend therapy sessions at least once per week.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-04; Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Watkins, Ph.D., Principal Investigator — Duke University; Jean C. Beckham, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LoSavio ST, Beckham JC, Wells SY, Resick PA, Sherwood A, Coffman CJ, Kirby AC, Beaver TA, Dennis MF, Watkins LL. The effect of reducing posttraumatic stress disorder symptoms on cardiovascular risk: Design and methodology of a randomized clinical trial. Contemp Clin Trials. 2021 Mar;102:106269. doi: 10.1016/j.cct.2021.106269. Epub 2021 Jan 8. PMID 33429088

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total protocol enrollment was 112. Participants assigned to the Waitlist Period Control group were given the option to receive Cognitive Processing Therapy (CPT) after their second assessment. 27 of the 34 control group participants opted to receive CPT.
Groups:
- CPT-C After WP-CON: Any participant assigned to the WP-CON group will be given the opportunity to receive CPT-C after the post-waiting period assessment. Participants are not required to participate in this therapy or the study assessments; it is completely voluntary. Any data collected from this group of participants will not be included in primary or secondary outcome analysis.
Period: Main Study
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON) | CPT-C After WP-CON
Started | 78 | 34 | 0
Completed | 70 | 32 | 0
Not Completed | 8 | 2 | 0
Not completed — Lost to Follow-up | 7 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: Optional Cross-Over
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON) | CPT-C After WP-CON
Started | 0 | 0 | 27
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON) | Total
Number analyzed (Participants) | 78 | 34 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.59 (6.78) | 52.68 (6.34) | 51.92 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 19 | 63
  Male | 34 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 76 | 33 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 23 | 68
  White | 26 | 9 | 35
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 34 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post-Intervention in 24-hour Heart Rate Variability (HRV) Estimated From the Standard Deviation of the Interbeat Interval of Normal Sinus Beats (SDNN)
Description: 24-hour HRV measured from SDNN was obtained from 24-hours of ambulatory electocardiograph (ECG) recordings. Inclusion criteria for HRV requires that at least 80% of the recording show normal sinus rhythm. SDNN is an independent predictor of coronary heart disease and cardiac death. Means for SDNN are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: At baseline in the CPT group, 3 participants had unusable HRV based on HRV inclusion criteria and 1 participant had an allergic reaction requiring early removal of the recorder. Imputation was used to impute outcomes for the post-intervention missing data (11 drop-outs (9 in the CPT group and 2 in the WP-CON group) and 2 additional participants in the CPT refused to wear the recorder post-intervention (one of which experienced the allergic reaction at baseline).
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 74 | 34
milliseconds
  Baseline | 118 (42) | 113 (38)
  Post-intervention | 123 (45) | 108 (36)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [-2.7 to 22.3]

2. Secondary Outcome: Change From Baseline to Post-Intervention in 24-hour Heart Rate Variability (HRV) Estimated From Low Frequency HRV (LF-HRV)
Description: 24-hour HRV measured from LF-HRV was obtained from 24-hours of ambulatory electrocardiograph (ECG) recordings. Inclusion criteria for HRV requires that at least 80% of the recording show normal sinus rhythm. LF-HRV is a frequency domain measure of HRV which captures all heart rate variations occurring over the frequency band linked to sympathetic vasomotor oscillations. Higher LF-HRV reflects stronger baroreflex cardiovascular control which is offset by increases in cardiac efferent sympathetic activity during periods of acute stress and physical activity. Low levels of LF-HRV are predictive of incident diabetes and increased coronary heart disease risk. Means for LF-HRV are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln msec2
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 74 | 34
ln msec2
  Baseline | 5.9 (1.1) | 5.9 (1.0)
  Post-intervention | 5.9 (1.1) | 5.7 (1.0)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5]

3. Secondary Outcome: Change in Heart Rate Variability (HRV) Measured by Holter Monitor, as Indicated by High Frequency HRV (HF-HRV)
Description: 24-hour HRV measured from HF-HRV was obtained from 24-hours of ambulatory electocardiograph (ECG) recordings. Inclusion criteria for HRV requires that at least 80% of the recording show normal sinus rhythm. HF-HRV is a frequency domain measure of HRV which captures all heart rate variations occurring over the frequency band linked to respiration. Higher HF-HRV reflects stronger parasympathetic cardiac control. Low levels of HF-HRV are predictive of increased coronary heart disease risk. Means for HF-HRV are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln msec2
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 74 | 34
ln msec2
  Baseline | 4.9 (1.1) | 5.0 (1.1)
  Post-intervention | 5.0 (1.1) | 4.8 (1.1)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.027, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.0 to 0.6]

4. Secondary Outcome: Change in Heart Rate Variability (HRV) as Measured by Root Square Mean of Successive Interbeat Interval Differences (RMSSD)
Description: 24-hour HRV measured from RMSSD was obtained from 24-hours of ambulatory electocardiograph (ECG) recordings. Inclusion criteria for HRV requires that at least 80% of the recording show normal sinus rhythm. RMSSD is a time domain measure of HRV which captures heart rate variations occurring over the frequency band linked to respiration. Higher RMSSD reflects stronger parasympathetic cardiac control. Means for RMSSD are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 74 | 34
milliseconds
  Baseline | 23.3 (9.9) | 24.7 (12.5)
  6-week follow-up | 24.3 (12.9) | 22.1 (10.8)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [0.5 to 7.1]

5. Secondary Outcome: Change From Baseline to Post-Intervention in 24-hour Urinary Excretion of Norepinephrine
Description: 24-hour urinary excretion of norepinephrine was obtained from 24-hours of urine collection. Inclusion criteria for 24-hour urine collection requires that at least 300 milliliters of urine be collected. Norepinephrine levels have been found to be elevated in PTSD and following trauma exposure. Norepinephrine is implicated in the association between cardiovascular disease and stress. Means for norepinephrine are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: At baseline in the WP-CON group, 1 participant had unusable urinary norepinephrine based on the 24-hour urine inclusion criteria. Imputation was used to impute the missing data from the the 14 participants who did not have post-intervention data either due to dropping out of the study (8 in the CPT group and 2 in the WP-CON group), due to technical problems with sample analysis (n=2), failure to meet inclusion criteria for urine collection (n=1) or refusal to collect urine (n=1)
Measure: Mean (Standard Deviation); unit: nanograms per milligram
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 78 | 33
nanograms per milligram
  Baseline | 36.3 (16.0) | 39.8 (22.8)
  Post-intervention | 33.6 (15.0) | 38.6 (17.4)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-9.8 to 2.0]

6. Secondary Outcome: Change From Baseline to Post-Intervention in 24-hour Urinary Excretion of Epinephrine
Description: 24-hour urinary excretion of epinephrine was obtained from 24-hours of urine collection. Inclusion criteria for 24-hour urine collection requires that at least 300 milliliters of urine be collected. Epinephrine levels have been found to be elevated in PTSD and following trauma exposure. Epinephrine is implicated in the association between cardiovascular disease and stress. Means for epinephrine are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: At baseline in the WP-CON group, 1 participant had unusable urinary norepinephrine based on the 24-hour urine inclusion criteria. Imputation was used to impute the missing data from the 14 participants who did not have post-intervention data due to either dropping out of the study (8 in the CPT group and 2 in the WP-CON group), due to technical problems with sample analysis (n=2), failure to meet inclusion criteria for urine collection (n=1) or refusal to collect urine (n=1)
Measure: Mean (Standard Deviation); unit: nanograms per milligram
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 78 | 33
nanograms per milligram
  Baseline | 4.4 (3.2) | 5.0 (3.5)
  Post-intervention | 3.3 (2.1) | 3.9 (2.0)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.3 to 0.4]

7. Secondary Outcome: Change From Baseline to Post-Intervention in High Sensitivity C-Reactive Protein (Hs-CRP)
Description: Peripheral inflammation was measured from fasting levels of CRP. Inclusion criteria for measurement of hsCRP requires that the participant be free from active infections or acute inflammatory conditions; therefore, participants were required to be free of fever, infections, and acute inflammatory conditions for a minimum of 7 days prior to the blood draw. Oral temperatures were obtained from all participants to check for sickness at the time of blood draw. CRP will be measured because it has a strong correlation with cardiovascular morbidity and mortality. Means for hs-CRP are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: At baseline in the CPT group, 3 participants reported infections which violated protocol criteria and 1 sample was not analyzed due to technical problems. At baseline in the WP-CON group, 1 participant refused blood draw. Imputation was used to impute the missing data from the 17 participants who either dropped out (9 in the CPT group and 2 in the WL-CON group), had infection (1 in the CPT group), experienced technical problems (4 in the CPT group), or refused (1 in the WP-CON group)
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 74 | 33
milligrams per liter
  Baseline | 4.0 (6.4) | 3.6 (3.7)
  Post-intervention | 3.9 (5.8) | 3.9 (5.8)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.86, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.8 to 1.5]

8. Secondary Outcome: Change From Baseline to Post-Intervention in Flow-Mediated Dilation (FMD)
Description: Vascular endothelial function was measured under fasting conditions from the percent change in dilation of the brachial artery following controlled occlusion of the artery. FMD is a measure of health of blood vessels. Lower flow mediated dilation is associated with poor cardiovascular health. FMD was measured because it has been correlated with cardiovascular morbidity and mortality and is reduced following trauma exposure. Means for FMD are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: Imputation was used to impute data from the 11 participants who were missing post-intervention data due to dropping out of the study (9 in the CPT group and 2 in the WL-CON group).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 78 | 34
percent change
  Baseline | 2.5 (3.4) | 3.6 (3.8)
  Post-intervention | 3.4 (3.9) | 3.7 (4.2)
Statistical Analysis 1: Comparison: Cognitive Processing Therapy - Cognitive vs Waiting Period Control (WP-CON); This is the analysis of between-group difference in change from baseline to 6-week follow-up; Test type: Superiority; p = 0.77, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.7 to 1.2]

9. Post Hoc Outcome: Change From Baseline to Post-Intervention in Fasting Plasma Insulin
Description: Fasting plasma insulin is a measure of insulin resistance and is a independent predictor of cardiovascular mortality and of autonomic neuropathy. PTSD has been associated with increased incidence of diabetes and metabolic dysfunction. Means for fasting insulin are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: Subgroup of participants with no history of diabetes.
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 61 | 26
uIU/mL
  Baseline | 15.4 (13.2) | 14.0 (9.4)
  Post-intervention | 11.6 (7.0) | 19.3 (17.5)

10. Post Hoc Outcome: Change From Baseline to Post-Intervention in Fasting Plasma Glucose
Description: Fasting plasma glucose is a measure of diabetes risk and is a independent predictor of cardiovascular mortality and of autonomic neuropathy. PTSD has been associated with increased incidence of diabetes and metabolic dysfunction. Means for fasting glucose are listed below, and evaluation of change in scores can be found in statistical analysis 1.
Time Frame: Baseline & post-intervention (up to 20 weeks)
Population: Subgroup of participants with no history of diabetes.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON)
Number analyzed (Participants) | 61 | 26
mg/dL
  Baseline | 88.3 (12.0) | 87.7 (12.0)
  Post-intervention | 88.2 (13.3) | 90.9 (13.2)

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Arm/Group | Cognitive Processing Therapy - Cognitive | Waiting Period Control (WP-CON) | CPT-C After WP-CON
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/34 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/34 | 0/27
Other Adverse Events (participants affected / at risk) | 13/78 | 6/34 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Processing Therapy - Cognitive (N=78) | Waiting Period Control (WP-CON) (N=34) | CPT-C After WP-CON (N=27)
hospitalization due to self-harm (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Pt. was hospitalized overnight after cutting herself. Pt. had a pre-existing history of nonsuicidal self injury.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Processing Therapy - Cognitive (N=78) | Waiting Period Control (WP-CON) (N=34) | CPT-C After WP-CON (N=27)
increased depression or anxiety (Psychiatric disorders) | 7 (9) | 2 (2) | 3 (3)
skin rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 0 (0) — Related to wearing electrodes
nausea and lightheadedness due to fasting (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02736929/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT02736929/ICF_001.pdf